CLINICAL TRIAL: NCT03158220
Title: An Open-Label Phase III Clinical Trial to Study the Immunogenicity and Tolerability of GARDASIL®9 (A Multivalent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] Vaccine) in Adult Women (27- to 45-Year-Olds) Compared to Young Adult Women (16 to 26 Year Olds)
Brief Title: Immunogenicity and Tolerability of Broad Spectrum Human Papillomavirus (HPV) Vaccine in Adult and Young Adult Women (V503-004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-004
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult Women 27- to 45-years Old (Experimental): Adult women 27- to 45-years old will receive V503 vaccination, 0.5 mL in a 3-dose regimen administered on Day 1, Month 2, and Month 6.
  Interventions: Biological: V503
- Young Adult Women 16- to 26-years Old (Active Comparator): Young adult women 16- to 26-years old will receive V503 vaccination, 0.5 mL in a 3-dose regimen administered on Day 1, Month 2, and Month 6.
  Interventions: Biological: V503

INTERVENTIONS:
Biological: V503 — V503 vaccination, 0.5 mL in a 3-dose regimen administered on Day 1, Month 2, and Month 6
  Other Names: GARDASIL®9 (HPV 9-valent vaccine [recombinant, adsorbed]); HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58

SUMMARY:
This study will assess the safety and immunogenicity of GARDASIL®9 (V503) in 16- to 45-year-old women. The primary hypothesis of the study states that anti-HPV 16, 18, 31, 33, 45, 52, and 58 geometric mean titers (GMTs) at 4 weeks postdose 3 are non-inferior in adult women as compared with GMTs in young adult women.

ELIGIBILITY:
Inclusion Criteria:

* good physical health

Exclusion Criteria:

* history of an abnormal Pap (Papanicolaou) test or abnormal cervical biopsy results
* history of HPV-related condition
* history of known prior vaccination with an HPV vaccine
* pregnant
* user of recreational or illicit drugs
* history of severe allergic reaction, including known allergy to any vaccine component
* immunocompromised
* history of certain medications or is currently taking or has taken certain medications (details will be discussed at the time of consent)
* has thrombocytopenia or other coagulation disorder
* concurrently enrolled in a clinical study of investigational agent

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1212 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- Austria (2):
  - Universitatsklinik fuer Frauenheilkunde und Geburtshilfe ( Site 0002), Graz
  - Klin. Abtlg. fuer Gynaekologie und Geburtshilfe ( Site 0001), Vienna
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen ( Site 0007), Edegem
  - Universitair Ziekenhuis Gent ( Site 0006), Ghent
  - Universitair Ziekenhuis Gasthuisberg ( Site 0005), Leuven
  - University of Antwerp ( Site 0004), Wilrijk
- Finland (5):
  - HUS Katiloopiston sairaala ( Site 0009), Helsinki
  - Ita-Helsingin Rokotetutkimuskeskus ( Site 0011), Helsinki
  - Porin Rokotetutkimusklinikka ( Site 0012), Pori
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0010), Tampere
  - Turun rokotetutkimusklinikka ( Site 0037), Turku
- Germany (5):
  - Universitaetsmedizin Berlin Charite ( Site 0016), Berlin
  - Universitaetsklinikum Duesseldorf ( Site 0014), Düsseldorf
  - Praxis Dr. Peters ( Site 0015), Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0017), Hamburg
  - Universitaetsklinikum Tuebingen ( Site 0013), Tübingen
- Italy (3):
  - Istituto Nazionale dei tumori ( Site 0020), Milan, Milan
  - Ospedale San Raffaele ( Site 0022), Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello ( Site 0023), Palermo
- Spain (5):
  - CAP Centelles ( Site 0027), Centelles, Barcelona
  - Complejo Hospitalario de Torrecardenas ( Site 0030), Almería
  - Institut Catala Oncologia de Bellvitge - ICO ( Site 0026), L'Hospitalet de Llobregat
  - Hospital Sanitas La Moraleja ( Site 0031), Madrid
  - Hospital Universitario Infanta Leonor ( Site 0028), Madrid

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Joura EA, Ulied A, Vandermeulen C, Rua Figueroa M, Seppa I, Hernandez Aguado JJ, Ahonen A, Reich O, Virta M, Perino A, Peris Tuser M, Peters K, Origoni M, Raspagliesi F, Tjalma WAA, Tummers P, Woelber L, Nieminen P, van Damme P, Sehouli J, Fiol Ruiz G, Brucker S, Fehm T, Cheon K, Rawat S, Luxembourg A, Wittke F. Immunogenicity and safety of a nine-valent human papillomavirus vaccine in women 27-45 years of age compared to women 16-26 years of age: An open-label phase 3 study. Vaccine. 2021 May 12;39(20):2800-2809. doi: 10.1016/j.vaccine.2021.01.074. Epub 2021 Mar 3. PMID 33676783

RESULTS

PARTICIPANT FLOW:
Groups:
- Women 16-26 Years of Age: Young adult women 16- to 26-years old received V503 vaccination, 0.5 mL in a 3-dose regimen administered on Day 1, Month 2, and Month 6.
- Women 27-45 Years of Age: Adult women 27- to 45-years old received V503 vaccination, 0.5 mL in a 3-dose regimen administered on Day 1, Month 2, and Month 6.
Period: Overall Study
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Started | 570 | 642
Vaccination 1 | 570 | 640
Vaccination 2 | 563 | 635
Vaccination 3 | 556 | 629
Completed | 553 | 626
Not Completed | 17 | 16
Not completed — Screen Failure | 0 | 1
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Status unknown | 0 | 1
Not completed — Lost to Follow-up | 8 | 5
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age | Total
Number analyzed (Participants) | 570 | 642 | 1212
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (2.8) | 35.8 (5.5) | 29.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 570 | 642 | 1212
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 21 | 7 | 28
  Not Hispanic | 548 | 634 | 1182
  Unknown | 1 | 1 | 2
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 17 | 10 | 27
  Black or African American | 5 | 3 | 8
  Multiple | 7 | 1 | 8
  White | 539 | 627 | 1166

OUTCOME MEASURES:

1. Primary Outcome: Anti-HPV Geometric Mean Titers (GMTs) for Each Anti-HPV Type
Description: Antibodies to the HPV types contained in V503 were measured using a competitive luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL). Statistical comparisons between arms was performed for the HPV types considered oncogenic (HPV Types 16/18/31/33/45/52/58).
Time Frame: 4 weeks post vaccination 3 (Month 7)
Population: Received all 3 vaccinations of the correct dose and within acceptable day ranges, had evaluable serology results at Day 1 and Month 7, must have been seronegative to the appropriate HPV type at Day 1 and had no protocol deviations that could interfere with the evaluation of participant's immune response to the 9vHPV vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 485 | 533
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 421 | 448
  Anti-HPV 6 | 787.8 [732.5 to 847.2] | 638.4 [594.9 to 685.0]
  Anti-HPV 11: number analyzed (Participants) | 421 | 448
  Anti-HPV 11 | 598.7 [558.7 to 641.6] | 453.5 [424.1 to 485.0]
  Anti-HPV 16: number analyzed (Participants) | 436 | 448
  Anti-HPV 16 | 3075.8 [2863.4 to 3303.9] | 2147.5 [2001.1 to 2304.5]
  Anti-HPV 18: number analyzed (Participants) | 421 | 471
  Anti-HPV 18 | 744.5 [685.0 to 809.1] | 532.1 [491.8 to 575.7]
  Anti-HPV 31: number analyzed (Participants) | 447 | 488
  Anti-HPV 31 | 596.1 [551.1 to 644.9] | 395.7 [367.0 to 426.6]
  Anti-HPV 33: number analyzed (Participants) | 457 | 493
  Anti-HPV 33 | 354.5 [331.7 to 378.9] | 259.0 [242.9 to 276.1]
  Anti-HPV 45: number analyzed (Participants) | 470 | 515
  Anti-HPV 45 | 214.9 [197.7 to 233.7] | 145.6 [134.4 to 157.7]
  Anti-HPV 52: number analyzed (Participants) | 456 | 496
  Anti-HPV 52 | 346.5 [324.0 to 370.5] | 244.7 [229.4 to 261.0]
  Anti-HPV 58: number analyzed (Participants) | 451 | 478
  Anti-HPV 58 | 428.0 [399.4 to 458.6] | 296.4 [277.1 to 317.0]
Statistical Analysis 1: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 16; Test type: Non-Inferiority — Non-inferiority of GMT in 27-45 year-olds relative to 16-26 year-olds was demonstrated if the lower limit of the 95% confidence interval (CI) for the fold difference was greater than 0.5; p < 0.001, ANOVA — Analysis of variance (ANOVA) model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.70, 95% CI 2-sided [0.63 to 0.77] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 2: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 18; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — Analysis of variance (ANOVA) model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.71, 95% CI 2-sided [0.64 to 0.80] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 3: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 31; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — ANOVA model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.66, 95% CI 2-sided [0.60 to 0.74] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 4: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 33; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — ANOVA model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.73, 95% CI 2-sided [0.67 to 0.80] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 5: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 45; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — ANOVA model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.68, 95% CI 2-sided [0.60 to 0.76] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 6: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 52; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — ANOVA model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.71, 95% CI 2-sided [0.64 to 0.78] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds
Statistical Analysis 7: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Anti HPV 58; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — ANOVA model with response of log individual titers and a fixed effect for age groups; Fold Difference = 0.69, 95% CI 2-sided [0.63 to 0.76] — Fold difference calculated as GMT 27-45 year-olds/GMT 16-26 year-olds

2. Secondary Outcome: Percentage of Participants That Experienced at Least 1 Adverse Event (AE)
Description: An AE is any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants with 1 or more AEs was assessed.
Time Frame: Up to 1 month post vaccination 3 (up to 7 months)
Population: All participants that received at least 1 vaccination and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 570 | 640
Percentage of Participants | 92.8 | 92.5

3. Secondary Outcome: Percentage of Participants Who Had Study Vaccine Discontinued Due to Adverse Event.
Description: An adverse event is any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The percentage of participants who discontinued the study vaccine due to an adverse event regardless of study completion status was assessed.
Time Frame: Up to 1 month post vaccination 3 (up to 7 months)
Population: All participants that received at least 1 vaccination and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 570 | 640
Percentage of Participants | 0.0 | 0.2

4. Secondary Outcome: Percentage of Participants With at Least 1 Solicited Injection-site Adverse Event
Description: Participants were asked to record any injection-site reactions prompted in the Vaccination Report Card, i.e., injection-site tenderness, swelling, or redness, occurring after each study vaccination (solicited injection-site reactions). The percentage of participants with 1 or more solicited injection-site AE was assessed.
Time Frame: Up to 5 days post any vaccination
Population: All participants that received at least 1 vaccination and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 570 | 640
Percentage of Participants | 87.2 | 84.7
Statistical Analysis 1: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Test type: Other; p = 0.212, Miettinen & Nurminen; Difference in Percentages = -2.5, 95% CI 2-sided [-6.4 to 1.4] — Difference in percentages calculated as % Women 27-45 Years of Age minus % Women 16-26 Years of Age

5. Secondary Outcome: Percentage of Participants That Reported at Least 1 Systemic Adverse Event
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Systemic AEs are those not categorized as injection-site AEs. The percentage of participants that reported at least 1 systemic AE was assessed
Time Frame: Up to 15 days post any vaccination
Population: All participants that received at least 1 vaccination and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 570 | 640
Percentage of Participants | 66.3 | 64.4
Statistical Analysis 1: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Test type: Other; Difference in Percentages = -1.9, 95% CI 2-sided [-7.3 to 3.4] — Difference in percentages calculated as % Women 27-45 Years of Age minus % Women 16-26 Years of Age

6. Secondary Outcome: Percentage of Participants With Elevated Temperature (Fever)
Description: Participants were asked to record oral body temperature in the Vaccination Report Card. The percentage of participants with elevated temperature (≥37.8°C or 100.0°F) was assessed.
Time Frame: Up to 5 days post any vaccination
Population: All participants that received at least 1 vaccination and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 570 | 640
Percentage of Participants | 3.5 | 2.5
Statistical Analysis 1: Comparison: Women 16-26 Years of Age vs Women 27-45 Years of Age; Test type: Other; p = 0.300, Miettinen & Nurminen; Difference in Percentages = -1.0, 95% CI 2-sided [-3.1 to 0.9] — Difference in percentages calculated as % Women 27-45 Years of Age minus % Women 16-26 Years of Age

7. Secondary Outcome: Percentage of Participants Who Seroconverted to Each of the Anti-HPV Types
Description: Antibodies to the HPV types contained in V503 were measured using a competitive luminex immunoassay. The percentage of participants who were seronegative on Day 1 and have anti-HPV titer greater or equal to the type-specific serostatus cutoff at 4 weeks postdose 3 was assessed.
Time Frame: 4 weeks post vaccination 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
Number analyzed (Participants) | 485 | 533
Percentage of Participants
  Anti HPV 6: number analyzed (Participants) | 421 | 448
  Anti HPV 6 | 99.8 [98.7 to 100.0] | 100.0 [99.2 to 100.0]
  Anti HPV 11: number analyzed (Participants) | 421 | 448
  Anti HPV 11 | 100.0 [99.1 to 100.0] | 99.8 [98.8 to 100.0]
  Anti HPV 16: number analyzed (Participants) | 436 | 448
  Anti HPV 16 | 100.0 [99.2 to 100.0] | 100.0 [99.2 to 100.0]
  Anti HPV 18: number analyzed (Participants) | 421 | 471
  Anti HPV 18 | 100.0 [99.1 to 100.0] | 99.6 [98.5 to 99.9]
  Anti HPV 31: number analyzed (Participants) | 447 | 488
  Anti HPV 31 | 100.0 [99.2 to 100.0] | 99.8 [98.9 to 100.0]
  Anti HPV 33: number analyzed (Participants) | 457 | 493
  Anti HPV 33 | 100.0 [99.2 to 100.0] | 99.8 [98.9 to 100.0]
  Anti HPV 45: number analyzed (Participants) | 470 | 515
  Anti HPV 45 | 99.6 [98.5 to 99.9] | 99.2 [98.0 to 99.8]
  Anti HPV 52: number analyzed (Participants) | 456 | 496
  Anti HPV 52 | 100.0 [99.2 to 100.0] | 100.0 [99.3 to 100.0]
  Anti HPV 58: number analyzed (Participants) | 451 | 478
  Anti HPV 58 | 100.0 [99.2 to 100.0] | 99.8 [98.8 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to 1 month post vaccination 3 (up to 7 months)
Description: Population included all participants that received at least 1 vaccination.
Arm/Group | Women 16-26 Years of Age | Women 27-45 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/570 | 0/640
Serious Adverse Events (participants affected / at risk) | 6/570 | 8/640
Other Adverse Events (participants affected / at risk) | 518/570 | 574/640
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women 16-26 Years of Age (N=570) | Women 27-45 Years of Age (N=640)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basilar migraine (Nervous system disorders) | 0 (0) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women 16-26 Years of Age (N=570) | Women 27-45 Years of Age (N=640)
Nausea (Gastrointestinal disorders) | 31 (35) | 27 (32)
Fatigue (General disorders) | 28 (36) | 33 (42)
Injection site erythema (General disorders) | 112 (166) | 111 (163)
Injection site pain (General disorders) | 492 (1246) | 532 (1244)
Injection site swelling (General disorders) | 137 (206) | 152 (224)
Pyrexia (General disorders) | 36 (40) | 28 (31)
Nasopharyngitis (Infections and infestations) | 53 (57) | 56 (69)
Headache (Nervous system disorders) | 185 (297) | 200 (320)
Dysmenorrhoea (Reproductive system and breast disorders) | 51 (65) | 22 (27)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40 (44) | 46 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03158220/Prot_SAP_000.pdf